CLINICAL TRIAL: NCT05818384
Title: Wakaya: Rising Up for Choctaw Youth Health
Acronym: Wakaya
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michelle Johnson-Jennings, Professor, School of Social Work, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00015208; 1R01DA056416 (NIH)
Record Dates: First submitted 2023-03-27; First posted 2023-04-18 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-02

CONDITIONS: Obesity, Adolescent; Healthy Nutrition; Sedentary Behavior; Drug Abuse
Keywords: Native Americans; Youth; Oklahoma; Adolescents; Obesity prevention
MeSH Terms: conditions — Pediatric Obesity; Sedentary Behavior; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wait List Control (Experimental): Participants in the Wait List group will be randomly assigned to start the intervention 3 months later in the Summer.
  Interventions: Behavioral: Wakaya: Rising Up for Choctaw Youth Curriculum
- Wakaya (Immediate Group) (Experimental): Participants in the immediate group will be randomly assigned to start the intervention immediately in the Spring.
  Interventions: Behavioral: Wakaya: Rising Up for Choctaw Youth Curriculum

INTERVENTIONS:
Behavioral: Wakaya: Rising Up for Choctaw Youth Curriculum — An experiential, outdoor, nature-based program grounded in Choctaw values. It is a multi-level intervention that increases individual motivation and leadership skills to make healthy behavioral choices for behavior and exercise.

SUMMARY:
Investigators will conduct a two-group randomized waitlist-control trial to assess the efficacy of the Wakaya: Rising Up for Choctaw Youth Health program on improving physical activity, reducing sedentary behaviors and improving healthful eating habits as well as delaying or reducing alcohol, tobacco and other drug use. Wakaya is an experiential, outdoor, nature-based program grounded in Choctaw values. It is a multi-level intervention that increases individual motivation and leadership skills to make healthy behavioral choices for behavior and exercise.

DETAILED DESCRIPTION:
Study participants will be recruited in staggered cohorts with those in each recruitment wave receiving individual-level random assignment to either immediate intervention or waitlist control (3 months wait to intervention) for a total of 176 Choctaw youth (ages 12-19 years) participating over 5 years.

Recruitment strategies:

The following Recruitment strategies will be used: posting flyers, posters and brochures in stores, community centers, and other locations identified by our community advisors; and posting flyers in the tribal newspaper, school newsletters, tribal gathering areas, tribal health fairs, pow wows, local boys and girls clubs, youth centers, other local news outlets, and on a study webpage.

Screening:

* Participants will mainly be screened in-person, some may be screened over phone using the same talking points.
* Youth who are screened out will be given a community resource list.
* If a person is eligible, but declines to participate, they will be given a brief one-item exit question regarding general reason for non-participation.
* Eligible youth who agree to participate will be asked to schedule their baseline assessment.

After consent or assent and parental permission are obtained, CNO study staff will set up the study laptop and headphones that the participant will use to enter their responses to the baseline computer-assisted questionnaire.

Assessments:

The baseline assessment consists of a brief physical health assessment and a computer-assisted behavioral health survey administered by study staff. Youth participants are required to take a non-invasive physical health assessment (BMI with portable digital weight scale and height measure), identify the age they began puberty (girls < 12 years old began menstruation; boys <14 when voice changed "a lot" will be classified as early puberty) and to use an accelerometer for 7 days after the baseline assessment. They will also be asked to run or walk for 12 minutes. The computer-assisted behavioral health survey will ask a series of questions and take under 45 minutes to complete.

The assessments will be conducted via Audio-Computer Assisted Self-Interviews (ACASI) programmed into study computers. Participants will complete 4 surveys: baseline, immediately after Trail of Tears Walk, a three-month follow up,and a six-month follow-up.

Intervention Schedule:

Month 1-3: Up to 20 group sessions on Choctaw history, traditions, cultural systems and health beliefs. Experiential, outdoor activities are incorporated to promote group cohesion, improve relational worldviews, and connectedness to nature and the environment. Examples include activities on an outdoor ropes course or increasing physical activity by walking or gardening. Fitbits will be given to participants and peers can choose to support each other to meet goals on a social media platform. Up to 3 individual Motivational Interviewing sessions to identify personal change goals and community leadership.

Month 2-3: Attend an Overnight Culture Camp to strengthen group cohesion and synthesize goals.

Month 3: Walk on the Choctaw Trail of Tears and visit ancient sites. Upon completion, make a commitment to conduct a community-wide event based on personal and leadership goals and Trail experience.

Months 4-12: Up to 6 group meetings to plan community leadership events related to obesity prevention, includes an individual MI booster session to revise their personal & community leadership goals, digital storytelling training, and a community Traditional Games Olympiad. Participants may create a story related to healthful food habits, obesity prevention and alcohol, tobacco and other drug use (ATOD).

Month 9: Share digital stories, community events, and participate in a leadership ceremony.

Post-intervention: Ripple Effect Mapping focus groups among 64 individuals. A random selection of 12 youth per region and 4 nonparticipant community stakeholders i.e., elders, leaders in the community.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in Choctaw Nation of Oklahoma (CNO)
* Live within CNO tribal region for 12 months

YES to one of the following:

* Consumed sweetened beverages or processed/fast food 2x or more per week; OR
* Engaged in excessive sitting or lying around (>540 min/day) or engage in small screen recreation (>2 hours/day); OR
* Physical activity - spend <60 minutes/day outdoors or <2.5 hrs per week in moderate or vigorous physical activity OR spend <60 minutes a day in moderate or vigorous intensity aerobic activity; OR
* Engage in any T.V., small screen/video game recreation (> 2 hours/day)

Exclusion Criteria:

* opioid/methamphetamine drug use (2 times or more in past month)
* allergic reactions to food (e.g. peanuts), plant (poison oak or ivy) or insects (e.g. bees, fire ants) that caused difficulty in breathing or necessitated hospitalization or caused an anaphylactic reaction
* disability that prevents student from walking or from engaging in exercise
* aggressive, violent, combative or inappropriate behaviors
* inability to follow directions
* psychotic symptoms

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity assessed by self-report | Baseline; Immediate post-intervention (month 3); 3 months post (month 6); and 6 months post-intervention (month 9)
  Assessed by the International Physical Activity Questionnaire-Short Form (IPAQ) for youth and young adults. Results can be reported in categories (low, moderate or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Change in physical activity intensity associated with movement, measured by accelerometer | Baseline and 6 months post-intervention (month 9)
  An actigraph accelerometer measures vertical acceleration in counts per minute. It will be worn for 7 days. Mean counts per minute are calculated by dividing the sum of activity counts for a valid day be the number of minutes of wear time in a day for all valid days. Greater number of counts per minute indicates higher physical activity intensity. Change in mean counts per minute from baseline at 9 months will be assessed.
Change in sedentary behaviors over time | Baseline; Immediate post-intervention (month 3); 3 months post (month 6); 6 months post-intervention (month 9)
  Measured by the Youth Leisure-time Sedentary Behavior Questionnaire (YLSBQ) adapted for Choctaw Youth
Change in food and beverage habits over time | Baseline; Immediate post-intervention (month 3); 3 months post (month 6); 6 months post-intervention (month 9)
  Assessed by the Youth Risk Behavior Surveillance System (YRBS) 2023.
Change in beverage habits over time | Baseline; post-intervention (month 3); 3 months post (month 6); 6 months post-intervention (month 9)
  Assessed by the Modified Healthy Home Survey (2005- Beverages). It assesses the number of sweetened drinks consumed per week.

SECONDARY OUTCOMES:
Body Mass Index (BMI) change | Baseline; Immediate post-intervention (month 3); 3 months post (month 6); 6 months post-intervention (month 9)
  Mean or percentage change in BMI from baseline. Weight (kg) and height (meters) will be combined to report BMI as kg/m^2.
Weight change assessed via digital scale | Baseline; Immediate post-intervention (month 3); 3 months post (month 6); 6 months post-intervention (month 9)
  Mean weight change (kg)
Change in food addiction | Baseline; Immediate post-intervention (month 3); 3 months post (month 6); 6 months post-intervention (month 9)
  The Yale Food Addiction Scale is a validated measure that has been developed to identify those who are most likely to be exhibiting markers of substance dependence with the consumption of high fat/high sugar foods. Food addiction (dichotomous) can be "diagnosed" when three symptoms and clinically significant impairment or distress are present. Continuous version of the scale ranges from 0 symptoms to 7 symptoms. Higher indicates more symptoms and worse dependence on high fat or high sugar foods.
Change in tobacco use frequency (non-ceremonial use) assessed by self-report | Baseline; Immediate post-intervention (month 3); 3 months post (month 6); 6 months post-intervention (month 9)
  Tobacco use frequency will be assessed by 5 items on a 7-level ordinal scale from the YRBS 2023. With higher responses, reflecting greater tobacco use.
Change in alcohol use over time | Baseline; Immediate post-intervention (month 3); 3 months post (month 6); 6 months post-intervention (month 9)
  Alcohol use (current use, binge drinking) assessed by the YRBS 2023.
Change in marijuana use over time | Baseline; Immediate post-intervention (month 3); 3 months post (month 6); 6 months post-intervention (month 9)
  Past 30 day marijuana use (smoking, vaping, edibles) assessed by the YRBS 2023.
Change in drug and alcohol refusal self-efficacy | Baseline; Immediate post-intervention (month 3) 3 months post (month 6); 6 months post-intervention (month 9)
  The Specific Event Drug and Alcohol Refusal Self-Efficacy (SEDARE) measure captures the perceived likelihood that youth will use drugs and alcohol in specific situations on a 3-point scale (Yes, No, Unsure). The SEDARE produces two scores ranging from 0 to 8. Higher scores reflect greater self-efficacy to refuse alcohol or drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Johnson-Jennings, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Choctaw Nation of Oklahoma, Durant, Oklahoma
  - University of Washington, IWRI, School of Social Work, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No